CLINICAL TRIAL: NCT05060458
Title: Increasing Insight in Spatial Neglect: Unraveling Its Longitudinal Interaction With Motor Function After Stroke
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Wim Saeys, Professor, Universiteit Antwerpen
Other Study IDs: D0011000
Record Dates: First submitted 2021-09-08; First posted 2021-09-29 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Spatial Neglect; Postural Control
Keywords: Stroke; Postural control; Spatial neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Goal: Various studies suggest a negative association between spatial neglect and motor outcomes after stroke (Barrett & Muzaffar 2014) (Kwakkel 2014). Our goal is to assess:

* The longitudinal interaction of the recovery of spatial neglect with the recovery of motor function and outcomes (such as paresis, sitting balance and standing balance)
* Whether the association is different across the different subtypes of spatial neglect (visuospatial/personal/ADL-related)
* The role of compensation strategies for balance control in patients with spatial neglect

To do so, we will perform a longitudinal cohort study in which we will repetitively assess post-stroke patients using a comprehensive assessment approach for both spatial neglect and motor outcomes. With regards to neglect, we will evaluate various aspects of both visuospatial and personal neglect. For motor outcomes, we will combine clinical and instrumented (biomechanical) assessment methods to evaluate post-stroke recovery of leg paresis, (sitting and standing) balance and gait.

DETAILED DESCRIPTION:
Spatial neglect is a post-stroke disorder characterized by impaired awareness for stimuli located on the contralesional side of space. This neglect results in problems with reporting, responding or orienting toward contralesional stimuli, which cannot be explained by sensory or motor impairments. It can be present after a right- or left-sided brain lesion but is more frequently present in right-sided brain lesions. Within the first 2 weeks post-stroke, it occurs in approximately 50% of patients. Spontaneous neurological recovery of neglect follows a natural logistic pattern of improvement within the first 12 to 14 weeks post-stroke. Afterward, the curve flattens and the severity remains merely invariant, leaving 40% of patients with initial neglect still with symptoms at 1 year post-stroke.

The high frequency and persistence of spatial neglect might have major consequences; indeed, various studies suggest a negative association between spatial neglect and post-stroke recovery of motor function and abilities. Apart from the seemingly suppressive influence of VSN on the recovery of upper-limb strength and synergy acquisition, lower limb motor recovery, balance and functional mobility might also be affected. However, the longitudinal interactions between spatial neglect and lower limb motor recovery are complex and only partially understood, owing to a lack of prospective cohort studies evaluating this. Additionally, also the association between spatial neglect and balance and functional mobility is currently unclear. A comprehensive overview is lacking, even though both balance and functional mobility are likely to be affected in these patients. Indeed, spatial neglect is characterised by a spatial (orientational) bias of attention. This bias might reflect a disruption in spatial information processing, which is a neural process incorporating sensory information from multiple modalities, resolving sensory ambiguity and integrating afferent and efferent information. A bias in this information processing might impede postural control and therefore also balance and mobility. However, whether spatial neglect and these motor outcomes are longitudinally associated, and whether such association is similar for the different spatial neglect subtypes, is still unknown.

Our goal is to assess:

* The longitudinal interaction of the recovery of spatial neglect with the recovery of motor function and outcomes (such as paresis, sitting balance and standing balance)
* Whether the association is different across the different subtypes of spatial neglect (visuospatial/personal/ADL-related)
* The role of compensation strategies for balance control in patients with spatial neglect

To do so, we will perform a longitudinal cohort study in which we will repetitively assess post-stroke patients using a comprehensive assessment approach for both spatial neglect and motor outcomes. With regards to neglect, we will evaluate various aspects of both visuospatial and personal neglect. For motor outcomes, we will combine clinical and instrumented (biomechanical) assessment methods to evaluate post-stroke recovery of leg paresis, (sitting and standing) balance and gait.

Recruitment: as early as possible after stroke on fixed time-points post-stroke as recommended by the Stroke Recovery and Rehabilitation Roundtable (internationally renowned field experts). We include patients at: ≤14 days, 3 weeks, or 5 weeks post-stroke. Inclusion in RevArte rehabilitation hospital, UZA, GZA St-Augustinus, GZA St-Vincentius and Reva Geel.

Outcome measures: include measures for spatial neglect, motor function and balance/mobility.

Data analysis: linear mixed models will be fitted to evaluate study results and therefore mean change over time.

ELIGIBILITY:
Inclusion Criteria:

* First-ever, MRI- or CT-confirmed, ischemic or hemorrhagic, anterior circulation stroke
* Age: 18 - 90 years
* Moderate to severe weakness of the lower limb at baseline (MI </=75)
* Pre-morbid independence in activities of daily living (mRS </=2) and gait (FAC >3)
* Able to communicate and comprehend
* Sufficient motivation to participate
* Provided a written informed consent

Exclusion Criteria:

* Other neurological condition affecting motor functions of the lower limbs
* Pre-existing musculoskeletal impairment severely affecting the gait pattern
* Medically unstable
* Non-corrected vision disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-ever stroke patients (inpatient or outpatient)
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Change in Rivermead Mobility Index | Change from <14 days to 3 weeks
  Change in functional balance and mobility. Score from 0 to 15. Higher score means better performance.
Change in Rivermead Mobility Index | Change from 3 weeks - 5 weeks
  Change in functional balance and mobility. Score from 0 to 15. Higher score means better performance.
Change in Rivermead Mobility Index | Change from 5 weeks - 8 weeks
  Change in functional balance and mobility. Score from 0 to 15. Higher score means better performance.
Change in Rivermead Mobility Index | Change from 8 weeks - 12 weeks
  Change in functional balance and mobility. Score from 0 to 15. Higher score means better performance.
Change in Broken Hearts Test | Change from <14 days to 3 weeks
  Change in cancellation task for visuospatial neglect
Change in Broken Hearts Test | Change from 3 weeks to 5 weeks
  Change in cancellation task for visuospatial neglect
Change in Broken Hearts Test | Change from 5 weeks to 8 weeks
  Change in cancellation task for visuospatial neglect
Change in Broken Hearts Test | Change from 8 weeks to 12 weeks
  Change in cancellation task for visuospatial neglect
Functional Ambulation Categories | Change from <14 days to 3 weeks
  Walking evaluation. Score from 0-5. Higher score means better performance.
Functional Ambulation Categories | Change from 3 weeks to 5 weeks
  Walking evaluation. Score from 0-5. Higher score means better performance.
Functional Ambulation Categories | Change from 5 weeks to 8 weeks
  Walking evaluation. Score from 0-5. Higher score means better performance.
Functional Ambulation Categories | Change from 8 weeks to 12 weeks
  Walking evaluation. Score from 0-5. Higher score means better performance.

SECONDARY OUTCOMES:
Trunk Control Test - item quiet sitting for 30 seconds | <14 days, 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Sitting, hands on lap, feet of the ground. Score from 0 to 2. Higher score means better performance.
Berg Balance Scale - item quiet standing for 2 minutes | <14 days, 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Ability to stand unsupported. Score from 0 to 4. Higher score means better performance.
Motricity index - lower limbs | <14 days, 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Strength of the hip flexors, knee extensors and dorsiflexors (paretic vs non paretic limb)
Fügl-Meyer Motor Assessment - lower limbs | <14 days, 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Selectivity of the paretic lower limb
5m walk test | <14 days, 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Walking speed
Line Bisection Test | 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Visuospatial neglect test
Visuospatial Search Time Test | 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Visuospatial neglect test
Fluff Test | 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Personal neglect test
Tactile extinction test | 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  Personal neglect test
Catherine Bergego Scale | 3 weeks, 5 weeks, 8 weeks, 12 weeks post-stroke
  ADL related neglect test

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Edegem
  - RevArte, Edegem
  - GZA Ziekenhuis - campus St Augustinus & Campus St Vincentius, Wilrijk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Embrechts E, Schroder J, Nijboer TCW, van der Waal C, Lafosse C, Truijen S, Saeys W. Does visuospatial neglect contribute to standing balance within the first 12 weeks post-stroke? A prospective longitudinal cohort study. BMC Neurol. 2024 Jan 22;24(1):37. doi: 10.1186/s12883-023-03475-1. PMID 38254026